CLINICAL TRIAL: NCT04992559
Title: A Phase II, Open-Label, Single-arm Study of Toripalimab As Consolidation Therapy After Postoperative Radiotherapy or Chemoradiotherapy in Patients With Head and Neck Squamous Cell Carcinomas (HNSCC)
Brief Title: A Study of Toripalimab as Consolidation Therapy After Postoperative Chemoradiotherapy in HNSCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Song Fan, MD, Associate Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-KY-039
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Head and Neck Squamous Cell Carcinomas
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab Arm (Experimental): Toripalimab consolidation therapy
  Interventions: Drug: Consolidation Toripalimab

INTERVENTIONS:
Drug: Consolidation Toripalimab — Toripalimab consolidation therapy after radiotherapy or chemoradiotherapy, 240mg IV, every 3 weeks, until progressive disease (PD), start new anti-cancer therapy, intolerable toxicity, withdraw informed consent or other conditions that require study treatment discontinuation. Toripalimab will be given at a maximum of 12 months.

SUMMARY:
This study is a phase II, open label, single-arm and exploratory clinical trial. The purpose of this study is to observe the efficacy and safety of consolidation immunotherapy with Toripalimab following postoperative radiotherapy or chemoradiotherapy for patients with locally advanced head and neck squamous cell carcinomas (HNSCC).

ELIGIBILITY:
Inclusion Criteria:

* Postoperative with adverse prognostic factors in patients with locally advanced head and neck squamous cell carcinoma.
* Have received postoperative adjuvant radiotherapy (chemo) therapy, and the end of the treatment is not more than 2 months.
* Greater than or equal to 18 and less than 70 years of age at time of study entry.
* ECOG performance status of 0 or 1.
* Measurable disease as per RECIST 1.1.
* Screening labs must meet the following criteria and must be obtained within 14 days prior to registration:

  1. Adequate hepatic and renal function as demonstrated by

     1. Serum creatinine < 1.5 X ULN or CrCl > 40mL/min (if using the Cockcroft-Gault formula below):

        * Males: Creatinine CL (mL/min) = (Weight (kg) x (140 - Age))/(72 x serum creatinine (mg/dL)）
        * Females: Creatinine CL (mL/min) = (Weight (kg) x (140 - Age))/(72 x serum creatinine (mg/dL))x 0.85
     2. AST/ALT ≤ 3 x ULN
     3. Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
  2. Adequate bone marrow function as demonstrated by:

     1. Absolute Neutrophil Count >1,500/µL
     2. Platelets > 100 X 103/µL
     3. Hemoglobin > 9.0 g/dL
* Women of reproductive potential should have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 7 days of study enrollment.
* Women of reproductive potential must use highly effective contraception methods to avoid pregnancy for 3 months after the last dose of study drugs; "women of reproductive potential" is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal; menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes; in addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL.
* Men of reproductive potential who are sexually active with women of reproductive potential must use any contraceptive method with a failure rate of less than 1% per year; men who are receiving the study medications will be instructed to adhere to contraception for 3 months after the last dose of study drugs; men who are azoospermic do not require contraception.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent within 4 weeks of the first dose of treatment or has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had another known invasive malignancy within the previous 5 years （With the exception of basal cell carcinoma of the skin, carcinoma in situ of the cervix, and papillary carcinoma of the thyroid, which has been cured）.
* If subject received major surgery for any other reason, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Active, known or suspected autoimmune disease.
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has received prior therapy with an anti-PD-1 antibody .
* A history of allergic reaction attributed to compounds of similar chemical or biologic composition to the treatment or other agents used in the study.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 23 weeks after the last dose of trial treatment.
* Has a known history of Human Immunodeficiency Virus (HIV) infection (HIV 1/2 antibodies).
* Has known active Hepatitis B or C.
* Known history of active TB ( bacillus tuberculosis ).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2021-06-22 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
2-year Disease-Free Survival Rate | 2 years
  The 2-year DFS rate was defined as the rate of progression or death due to disease recurrence within 2 years.

SECONDARY OUTCOMES:
2-year overall survival rate | 2 years
  Number of patients with evidenced death / number of total patients.
Media Disease-free Survival (mDFS) | Up to 5 years
  The time at which disease progression or death due to disease progression occurred in 50% of patients.
Overall survival | 5 years
  Overall survival will be defined as the time from day 1 of study treatment until death from any cause.
Adverse events | 90 days after the first dose of study treatment
  Percentage of adverse events that are possibly, probably or definitely related to study treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong